CLINICAL TRIAL: NCT05820724
Title: Prostate Specific Membrane Antigen (PSMA) Scan and Multiparametric MRI for Prostate Biopsy Detection of Clinically Significant Prostate Cancer
Brief Title: PSMA PET Scan and mpMRI for Prostate Cancer Detection
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1685514-1
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer Diagnosis
Keywords: psma PETCT; prostate mpMRI; prostate needle biopsy; DCFPyL PET/CT
MeSH Terms: interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PSMA PET+mpMRI (Experimental): PSMA PET+mpMRI guided prostate biopsy
  Interventions: Diagnostic Test: PSMA PET scan; Drug: 18F- DCFPyl Injection
- mpMRI only (Active Comparator): mpMRI only guided prostate biopsy
  Interventions: Other: No PSMA PET

INTERVENTIONS:
Diagnostic Test: PSMA PET scan — Subjects will undergo DCFPyL PET/CT imaging and mpMRI imaging prior to the prostate biopsy. The decision for biopsy targets will be made based on the combination of the findings of mpMRI and PSMA scans. The intervention includes a mpMRI, a PSMA PET scan, and a prostate biopsy.
  Other Names: DCFPyL PET/CT imaging
  Arms: PSMA PET+mpMRI
Other: No PSMA PET — Subjects will undergo mpMRI imaging prior to the prostate biopsy. These subjects do not undergo a PSMA PET scan prior to the prostate biopsy. The decision for biopsy targets will be made based on the findings of mpMRI. The intervention includes a mpMRI and a prostate biopsy.
  Arms: mpMRI only
Drug: 18F- DCFPyl Injection — DCFPyL is a PSMA imaging ligand that was developed to enhance the detection of small lesions in the prostate or other pelvic areas. 18F- DCFPyl Injection will be administered prior to the PSMA PET/CT via an in-dwelling catheter placed in an antecubital vein or an equivalent venous access under the direct supervision of study personnel.
  Other Names: DCFPyl
  Arms: PSMA PET+mpMRI

SUMMARY:
Prospective, randomized, phase 2 clinical trial to determine if PSMA PET imaging plus mpMRI improves detection of clinically significant prostate cancer as compared to mpMRI alone.

DETAILED DESCRIPTION:
This a prospective, randomized, phase 2 clinical trial. We will enroll patients who underwent mpMRI of the prostate as part of their standard clinical care, have PI-RADS 4, or 5 lesion(s) on mpMRI, and are scheduled to undergo fusion guided prostate biopsy. Subjects that sign the consent form will be randomized to undergo DCFPyL PET/CT imaging or no PSMA PET imaging prior to the prostate biopsy. In the PSMA scan cohort, decision for biopsy targets will be made based on the combination of the findings of mpMRI and PSMA scans. In the no PSMA scan (control) group, the biopsy will be performed based on mpMRI findings. Each patient will undergo 12 core systematic biopsy as the standard of care. Two additional biopsies for each mpMRI and PSMA PET and overlap lesion will also performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PI-RADS 4-5 lesion(s) on mpMRI and have elected to undergo a prostate biopsy
* Prostate mpMRI completed within 9 months prior to enrollment
* Patient capable of providing written informed consent
* Patient willing to be randomized to prostate mpMRI only vs prostate mpMRI + DCFPyL PET/CT

Exclusion Criteria:

* Less than 18 years-old at the time of radiotracer administration
* Medical condition, serious concurrent illness, or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study procedures or compliance.
* Creatinine clearance exceeding institutional requirements for prostate mpMRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Detection of Clinically Significant Prostate Cancer | 12 weeks
  Percentage of mpMRI and PSMA PET lesions positive for clinically significant prostate cancer

SECONDARY OUTCOMES:
Detection of Clinically Insignificant Prostate Cancer | 12 weeks
  Percentage of mpMRI and PSMA PET lesions positive for clinically insignificant prostate cancer.
Difference in PSMA PET and mpMRI Clinically Significant Cancer Detection | 12 weeks
  Percentage of PSMA PET only (mpMRI negative) and PSMA PET overlapping with mpMRI lesions positive for clinically significant prostate cancer.
Correlation of PSMA PET intensity with Clinically Significant Prostate Cancer | 12 weeks
  Correlate intensity of PSMA PET lesions with clinically significant prostate cancer.
Correlation of AI Measures with Aggressiveness of Prostate Cancer | 12 weeks
  Correlate artificial intelligence measurement(s) (miPSMA index) of PSMA lesion(s) with aggressiveness of prostate cancer
Adverse Events Associated with 18F- DCFPyl | 12 weeks
  Safety - Patients will be monitored for adverse events during injection and for two hours after radiotracer administration.

CONTACTS AND LOCATIONS:
Overall Officials: William Aronson, MD, Principal Investigator — VA Greater Los Angeles Healthcare System
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No